CLINICAL TRIAL: NCT06691360
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of AK137 (Bispecific Antibody Targeting CD73 and LAG-3) in Patients With Advanced Malignant Tumors
Brief Title: AK137 (Bispecific Antibody Targeting CD73 and LAG-3) in Patients With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK137-101
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK137 (Experimental): Each subject will receive a single dose of AK137 every 3-week cycle (Q3W) or every 2-week cycle (Q2W). Participants may continue on study drug until unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: AK137

INTERVENTIONS:
Drug: AK137 — IV infusion, specified dose on specified days.

SUMMARY:
A Phase I open label, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and antitumor activity of AK137 in patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent.
2. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
3. Life expectancy ≥3 months.
4. Histologically or cytologically documented unresectable advanced or metastatic malignant tumor that has failed or intolerant of standard therapy, or for which no effective standard therapy is available.
5. Subject must have at least one measurable lesion according to RECIST Version1.1.
6. Adequate organ function.

Exclusion Criteria:

1. Any malignancy other than the disease under study within the past 3 years except for radically cured local cancers, such as basal cell skin cancer, carcinoma in situ of the cervix, or carcinoma in situ of breast.
2. Receipt of any anti-CD73, anti-LAG-3 treatment.
3. Experienced a toxicity that led to the permanent discontinuation of prior immunotherapy. All adverse events (AEs) while receiving prior immunotherapy have not completely resolved or resolved to Grade 1 prior to screening. Additionally, the use of immunosuppression other than corticosteroids was required.
4. Unresolved toxicities from prior anticancer therapy, defined as not having resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels specified in the inclusion/exclusion criteria, except for toxicities not considered a safety risk (e.g., alopecia, neuropathy, or asymptomatic laboratory abnormalities).
5. Major surgical procedure within 4 weeks prior to the first dose of AK137 or still recovering from prior surgery.
6. History of organ transplant.
7. Known allergy or reaction to any component of the AK137 formulation. History of severe hypersensitivity reactions to other mAbs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
AEs | From time ICF is signed until 90 days after last dose of AK137
  Incidence and severity of participants with adverse events
DLT | During the first 28-day of treatment with AK137

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
Disease Control Rate (DCR) | Up to approximately 2 years
Duration of Response (DoR) | Up to approximately 2 years
Time to response (TTR) | Up to approximately 2 years
Progression Free Survival (PFS) | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 2 years
Cmax of AK137 | From first dose of study drug through end of treatment (up to approximately 2 years)
Cmin of AK137 | From first dose of study drug through end of treatment (up to approximately 2 years)
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China